CLINICAL TRIAL: NCT01377662
Title: PHASE IIA: Randomized, Double Blind, Placebo Controlled, Single Center Clinical Trial of a Combination of a Novel Ondansetron Formulation (OND-PR002) and Immediate-Release Methylphenidate (Ritalin®)
Brief Title: PHASE IIA: Trial of a Novel Ondansetron Formulation (OND-PR002) and Immediate-Release Methylphenidate (Ritalin®)(OND003IND)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tong Lee (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor-Investigator, Tong Lee, Associate Professor Psychiatry and Behavorial Science, Duke University
Organization: Duke University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Pro00030921; 1RC2DA028905-01 (NIH)
Record Dates: First submitted 2011-06-12; First posted 2011-06-21 (Estimated); Last update posted 2014-10-07 (Estimated); Status verified 2014-09

CONDITIONS: Methamphetamine Dependence; Cocaine Dependence
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — Ondansetron; Methylphenidate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo: Two dextrose capsules for Ond-PR002 and MPh-IR
- OND-PR002 and MPh-IR (Experimental)
  Interventions: Drug: OND-PR002 and MPh-IR

INTERVENTIONS:
Drug: OND-PR002 and MPh-IR — Drug: OND-PR002
  Single daily oral doses of 8 mg Ond-PR002
  Drug: MPh-IR
  Single daily oral doses of 20 mg MPh-IR
  Other Names: Ondanasetron; Zofran®; Methylphenidate; Ritalin®
  Arms: OND-PR002 and MPh-IR
Other: Placebo: Two dextrose capsules for Ond-PR002 and MPh-IR — Single daily oral doses
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
The main purpose of this study is to determine the outcome of a drug combination treatment on detoxified and stabilized methamphetamine (METH) and/or cocaine (COC) dependent users. The combination regimen consists of oral administration of a generic immediate-release methylphenidate (MPh-IR) formulation (e.g., Ritalin®) and a novel delayed, pulsatile-release formulation of the antiemetic ondansetron (Ond-PR002). Various psychological assessment tools and functional magnetic resonance imaging (fMRI) will be used to assess the treatment outcome. In addition to the treatment outcome measures, we will determine whether the 14-day, once-a-day treatment leads to significant changes in the pharmacokinetic/pharmacodynamic (PK/PD), safety and tolerability parameters of MPh-IR and/or Ond-PR002 formulations and drug-drug interactions between the two drugs.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must give written informed consent.
* Detoxified METH/COC-dependent male and/or female subjects between 18 and 45.
* Females with Body Mass Index (BMI) of 18-36 kg/m2. Males with BMI of 20-36 kg/m2.
* Subjects in good health determined by screening examination.
* Subject must have adequate veins for intravenous site.
* Subjects must be mentally stable for minimum of 3 months.
* Non-clinically significant hematology clinical laboratory results.
* Subjects must have hematocrit of greater than or equal to 33%.
* Non-clinically significant screening 12-lead ECG and QT interval (time for ventricular depolarization and repolarization to occur) corrected by Fridericia formula (QTcF) of < 440 msec for male and < 460 msec for females.
* Subjects must be right-handed (control for handed-related differences) in lateralized patterns of brain function.
* Ability to identify visual cues during fMRI.
* Subjects' VAS score must be above 20.

Exclusion Criteria:

* Subjects who consume more than 28 units of alcohol per week.
* Subjects who test positive for drugs of abuse or alcohol.
* Current use of nicotine replacement therapy or other smoking cessation treatment.
* Use of other investigational drugs within 30 days, or at least 5 half-lives of a study medication prior to enrollment.
* Subjects being treated with other psychotropic drug will be excluded based on PI's clinical judgment and potential drug-drug adverse reactions with study drugs.
* Subjects on prescribed, over-the-counter (OTC) or nutraceutical drugs that may influence the PK, safety or efficacy profiles of MPh-IR and/or Ond-PR002 will be excluded, or receive a washout prior to study enrollment. Subjects on drugs or substances known to be strong inhibitors or strong inducers of CYP 3A4/5 enzymes (enzymes involved in the metabolism of xenobiotics) or P-glycoprotein (P-gp) will be excluded in a similar manner.
* Subjects with heart disease or uncontrolled high blood pressure.
* Donation of any blood or plasma in the last month, or donation of >500mL of blood within the 3 months preceding study drug administration.
* History of serious adverse reaction or allergies to any drug or any other products used in the study.
* Allergies or intolerance to any of the products used in this study.
* Subjects who have allergies to pork-derived medications or those that contain pork-derived products.
* Inability to give informed consent or high likelihood of being unable to complete the necessary confinement.
* Subjects deemed inappropriate for this study by the Principal Investigator.
* Subjects with a documented brain abnormality, history of unexplained loss of consciousness, seizures, history of unexplained syncope, or history of transient ischemic attack or stroke within the past 6 months.
* History of concurrent illness that required hospitalization within 14 days prior to Day 1 or a clinically significant illness within 4 weeks prior to Day 1.
* History of clinically significant cardiovascular illness within the past 6 months.
* History of clinically significant hepatic, renal, pulmonary, metabolic, endocrine, infectious, gastrointestinal, hematologic, oncologic, retinopathy, or other medical disorders.
* History of unstable psychiatric illness requiring hospitalization within previous 6 months.
* Subjects with history of glaucoma, color blindness or other uncorrected vision problem.
* Subjects with QTcF interval duration greater than or equal to 440 msec (males) or greater than or equal to 460 msec (females) obtained from the 12-lead ECG recorder's measurements on the screening ECG.
* Individuals with a major condition that would make fMRI participation unsafe or uncomfortable.
* Females who are pregnant, breast-feeding or plan on becoming pregnant.
* Subjects who have a hematocrit < 33% or hemoglobin < 12.0 g/dL.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2011-08; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Efficacy of combined Ond-PR002 and MPh-IR treatment | 15 days
  Efficacy of combined Ond-PR002 and MPh-IR treatment in reducing the Visual Analogue Scale (VAS), Cocaine Selective Severity Assessment (CSSA) and Amphetamine Cessation Symptom Assessment (ACSA) craving scores in abstinent METH/COC abusers. Changes in cue-reactivity and inhibitory control deficits will be also assessed using functional magnetic resonance imaging (fMRI).

SECONDARY OUTCOMES:
Safety of combined MPh-IR + Ond-PR002 treatment | 15 days
  Number of subjects with clinically significant changes in vital signs, electrocardiogram (ECG), hematology or chemistry panel measurements and number of subjects with self-reported or observed adverse events or serious adverse events will be recorded.
Changes in the PK parameters of Ond-PR002 PK after 14-day treatment | 15 days
  Standard PK parameters of Ond-PR002 (e.g., maximum serum concentrations, time to reach max. concentration, apparent volume of distribution, etc.) will be calculated based on the serum drug concentrations, and statistical differences between Day 1 and Day 14 will be determined.
Changes in the PK parameters of MPh-IR PK after 14-day treatment | 15 days
  Standard PK parameters of MPh-IR on Day 1 and Day 14 will be calculated and statistically compared as described for Ond-PR002.
Tolerability of combined MPh-IR + Ond-PR002 treatment | 15 days
  Number of subjects with clinically significant changes in vital signs, electrocardiogram (ECG), hematology or chemistry panel measurements and number of subjects with self-reported or observed adverse events or serious adverse events will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Robert J Noveck, MD,PhD, Principal Investigator — Duke Clinical Research Unit; Ashwin A Patkar, MD, Principal Investigator — Psychiatry and Behavioral Sciences; Tong Lee, MD, PhD, Principal Investigator — Associate Professor Psychiatry and Behavorial Science, Duke University Medical Center
Locations (3):
- United States (3):
  - Duke Addictions Clinic, Durham, North Carolina
  - Duke Clinical Research Unit, Durham, North Carolina
  - SouthLight, Raleigh, North Carolina